CLINICAL TRIAL: NCT04445870
Title: Oncology Care Pathway's Modifications Impact During COVID-19 Pandemic : the ONCOCARE-COV Study
Acronym: ONCOCARE-COV
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 2020Ao001*
Record Dates: First submitted 2020-06-23; First posted 2020-06-24 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Electronic Health Records

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: data record — Data record on registers without medical files

SUMMARY:
In december 2019, SARS-CoV2 and its clinical manifestations, COVID-19, appeared in China and caused a pandemic. It led decision makers to prioritize emergency and intensive care dedicated to infection management. Other conditions, such as cancer screening, diagnosis, and treatment, may have been delayed during the containment period. Consequences of this "distraction effect" are being.

DETAILED DESCRIPTION:
Quantitative monthly data were analyzed from January 1, 2019 to May 31, 2020 in two French tertiary care center (University Hospital and Godinot Cancer Institute in Reims) and in a third center in the French epicenter (Colmar hospital). Oncologic activity indicators were extracted using oncologic electronic file, International Statistical Classification of Diseases and Related Health Problems, Tenth Revision (ICD-10) and nation-wide procedure codes (CCAM). The monthly number of different steps of oncology care pathway (screening, diagnosis and treatment) were collected: faecal immunochemical testing (FIT), mammography, histopathological and biomolecular/genetics analysis, nuclear medicine imaging, oncogeriatric evaluations, multidisciplinary tumor board meetings and files reviewed by meeting including first presentations, given personalized care program, medical announcement and reformulation nursing consultations, inserted central venous catheters, chemotherapy prepared and administered in chemotherapy day care, carcinologic surgeries and radiotherapy courses.

ELIGIBILITY:
Inclusion Criteria:

* Every adult patient entering an oncology care pathway between 01/01/2019 and 31/12/2020

Exclusion Criteria:

* <18 yo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient entering an oncology care pathway
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
data record | from 01/01/2019 to 31/12/2020
  faecal immunochemical testing (FIT), mammography, histopathological and biomolecular/genetics analysis, nuclear medicine imaging, oncogeriatric evaluations, multidisciplinary tumor board meetings and files reviewed by meeting including first presentations, given personalized care program, medical announcement and reformulation nursing consultations, inserted central venous catheters, chemotherapy prepared and administered in chemotherapy day care, carcinologic surgeries and radiotherapy courses.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided